CLINICAL TRIAL: NCT02244983
Title: Falls Of Unknown Origin (FUKNO) - Are Morbidity and Mortality Predictable in Patients Presenting With Falls?
Acronym: FUKNO
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: FUKNO_Protokoll_17-07-14
Record Dates: First submitted 2014-08-18; First posted 2014-09-19 (Estimated); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Accidental Falls; Underlying Disease of Falls

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- EFAB 65: Patients presenting to the emergency department with falls, above 65 years of age. Patients History will be taken as well as a blood sample
  Interventions: Other: Patients History

INTERVENTIONS:
Other: Patients History — History taking and drawing of a blood sample

SUMMARY:
It is the investigators goal to identify the prevalence of underlying diseases, make disposition more rational, and establish risk stratification tools in elderly patients presenting with falls. Additionally, the outcome of standard care (clinical assessment only for disposition) will be compared with a new approach combining the standard of care with biomarker assisted disposition of elderly patients presenting with falls. Therefore the investigators are looking at the following points.

Emergency department work-up

1. Prevalence of underlying disease
2. Developing algorithms for initial assessment Disposition

a. Establishing biomarker enhanced disposition planning by using risk-stratification tools b. Comparing geriatric emergency assessment to standardized disposition planning

ELIGIBILITY:
Inclusion Criteria:

* All fall patients aged 65 years and older who presented to the emergency department giving written informed consent

Exclusion Criteria:

* Patients below 65 years
* Non-fall patients above 65 years
* or lack of informed consent by patients or proxies

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All fall patients aged 65 years and older who presented to the emergency department giving written informed consentent
Sampling Method: Non-Probability Sample
Enrollment: 587 (Actual)
Dates: Start 2014-11-12 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2021-12-02 (Actual)

PRIMARY OUTCOMES:
Mortality | 30 Days
  Data Collection via Case Report Form

SECONDARY OUTCOMES:
Acute Morbidity | 30 Days
  Data Collection via Case Report Form
Institutionalisation | 180 Days
  Data Collection via interview with general practitioner
Disposition | 30 Days
  Data collection via case report form
Mortality | 90 Days
  Data Collection via Case Report Form
Mortality | 180 Days
  Data Collection via Case Report Form
Mortality | 365 Days
  Data Collection via Case Report Form

CONTACTS AND LOCATIONS:
Overall Officials: Roland Bingisser, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (4):
- Charité Campus Benjamin Franklin, Berlin, Berlin, Germany
- Switzerland (3):
  - University Hospital Basel, Basel, Canton of Basel-City
  - Cantonal Hospital Baselland, Bruderholz, Basel
  - Cantonal Hospital Baselland, Liestal, Liestal

REFERENCES:
- [Derived] Terhalle L, Arntz L, Hoffmann F, Arnold I, Hafner L, Picking-Pitasch L, Zuppinger J, Delport Lehnen K, Leuppi J, Somasundaram R, Nickel CH, Bingisser R. Nonspecific stress biomarkers for mortality prediction in older emergency department patients presenting with falls: a prospective multicenter observational study. Intern Emerg Med. 2025 Mar;20(2):585-595. doi: 10.1007/s11739-024-03693-6. Epub 2024 Jul 3. PMID 38960969